CLINICAL TRIAL: NCT00582855
Title: A 4-week, Parallel-group, Randomized, Double-blind, Placebo-controlled, Adaptive Proof of Concept Study of AQW051 at up to Three Dose Levels for the Treatment of Patients With Findings Consistent With Mild Alzheimer's Disease (AD) or Amnestic Mild Cognitive Impairment (Amnestic MCI)
Brief Title: Effect of AQW051 in Patients With Memory Impairment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A2104
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Mild Alzheimer's Disease; Amnestic Mild Cognitive Impairment
Keywords: AQW051; Mild Alzheimer's disease; Amnestic Mild Cognitive Impairment
MeSH Terms: interventions — 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AQW051
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQW051
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will investigate AQW051 in patients with either mild Alzheimer's disease or amnestic mild cognitive impairment. The effect on cognitive impairment will be measure using validated computerized tests which measure cognitive function. This study will also explore the safety and tolerability of AQW051 in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Meet the diagnostic criteria for either amnestic mild cognitive impairment (amnestic MCI) or mild Alzheimer's Disease (AD).
* Structural brain scan within the last 6 months prior to randomization that indicates no other underlying disease, in particular no evidence for vascular pathology except for normal age-related white matter/incidental white matter changes which is normal for this age group.
* Daily contact with a primary caregiver/partner

Exclusion Criteria:

* Immune therapy targeting Alzheimer beta amyloid within the last 12 months
* Institutionalized
* Disability that may prevent completion of all study requirements (e.g., blindness, deafness, or communication difficulty)
* Reported use of tobacco products in the previous 3 months or have a urine cotinine level greater than 500 ng/ml
* Past medical history of clinically significant electrocardiogram (ECG) abnormalities or a family history (grandparents, parents, and siblings) of prolonged QT-interval syndrome
* History or current diagnosis of conditions specified in the protocol.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Validated computerized cognitive assessment scores | Througout the study

SECONDARY OUTCOMES:
Validated computerized cognitive assessment scores, the different scores from the Alzheimer's Disease Assessment Score-cognitive subscale (ADAS-Cog), Quality of Life-Alzheimer disease scale and the Disability Assessment for Dementia scale | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (12):
- Canada (3):
  - Novartis Investigator Site, Halifax
  - Novartis Investigator Site, Montreal
  - Novartis Investigator Site, Toronto
- South Africa (3):
  - Novartis Investigator Site, Bloemfontein
  - Novartis Investigator Site, George
  - Novartis Investigator Site, Port Elizabeth
- United Kingdom (6):
  - Novartis Investigator Site, Blackpool
  - Novartis Investigator Site, Epping
  - Novartis Investigator Site, Glasgow
  - Novartis Investigator Site, Manchester
  - Novartis Investigator Site, Southampton
  - Novartis Investigator Site, Swindon